CLINICAL TRIAL: NCT01682382
Title: Collection of Whole Blood Specimens and Buccal Swabs From Subjects Diagnosed With CNV AMD, Dry AMD, and Age-Matched Controls to Assess the Association of Genetic Variants in Complement Factor H With Risk of Progression to CNV.
Brief Title: Association of Macular Pigment Optical Density (MPOD) and Genetic Variants in Complement Factor H in Subjects With Choroidal Neovascular (CNV)
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-AMD-103
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Age-related Macular Degeneration; Choroidal Neovascular Age-related Macular Degeneration
Keywords: age-related macular degeneration; choroidal neovascular age-related macular degeneration; genetics; macular pigment optical density (MPOD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood and buccal cells will be analyzed. Remnant samples will be stored for future research in AMD.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- choroidal neovascular (CNV) AMD subjects: Subjects diagnosed with CNV (AREDS Grade 4b)
- dry AMD subjects: Subjects diagnosed with dry AMD (AREDS Grade 3)
- age-matched controls: Subjects without AMD (AREDS Grade 1)

SUMMARY:
Subjects with wet AMD, dry AMD, and age-matched controls will undergo routine occular measurements, will provide a blood and cheek cell sample, and will have macular pigment optical density (MPOD) measured to determine if there is an association between genetics, MPOD and the risk of progression to wet AMD.

ELIGIBILITY:
Inclusion Criteria:

* subject is diagnosed with either CNV, dry AMD or is an age-matched control
* self reported as non-Hispanic Caucasian
* 60 years of age or older
* provides signed and dated informed consent
* agrees to provide 10 mL of whole blood and two buccal swabs

Exclusion Criteria:

* previous donation under this protocol

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-Hispanic Caucasian subjects 60 years of age and older diagnosed with either CNV or dry AMD and a cohort of age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Association between a genetic variant in the CFH gene and risk of progression to CNV | Baseline
  DNA extracted from blood and buccal cells collected from subjects with either CNV, dry AMD, and age-matched controls will be analyzed to investigate a genetic variant in the CFH gene and its association with risk of progression to CNV

SECONDARY OUTCOMES:
Genetic correlation between MPOD and risk of progression to CNV | baseline
  DNA extracted from blood and buccal cells collected from subjects with either CNV, dry AMD, and age-matched controls will be analyzed to investigate the correlation between genetics, MPOD, and risk of progression to CNV

CONTACTS AND LOCATIONS:
Locations (1):
- Morris Eye Group, Encinitas, California, United States